CLINICAL TRIAL: NCT03480984
Title: A Comparison Between Continuous Versus Intermittent Bolus Infusion of Paravertebral Blocks for Thoracic Surgery: A Randomized Controlled Trial
Brief Title: Continuous Versus Intermittent Bolus Infusion of Paravertebral Blocks for Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elird Bojaxhi, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-009991
Record Dates: First submitted 2018-02-01; First posted 2018-03-29 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators will not have direct access to settings on the pump
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmed Intermittent Bolus (Active Comparator): 6 mL 0.2% ropivacaine hourly, starting on arrival to PACU, given via an hourly programmed bolus
  Interventions: Other: Programmed Intermittent Bolus
- Continuous Infusion (Active Comparator): 6 mL 0.2% ropivacaine hourly, starting on arrival to PACU, given via continuous infusion
  Interventions: Other: Continuous Infusion

INTERVENTIONS:
Other: Programmed Intermittent Bolus — 6 mL 0.2% ropivacaine hourly, starting on arrival to PACU, given via an hourly programmed bolus
  Arms: Programmed Intermittent Bolus
Other: Continuous Infusion — 6 mL 0.2% ropivacaine hourly, starting on arrival to PACU, given via continuous infusion
  Arms: Continuous Infusion

SUMMARY:
The researchers are trying to determine pain medication consumption in the first 24 hours after surgery in patients given the standard continuous infusion of local anesthetic versus patients given the same total dose via programmed intermittent dosing. Both groups will receive the option of patient controlled pain medication as well as the same dose of pre-programmed pain medication. The only difference is the rate of administration: continuous vs. hourly intervals.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of planned thoracic surgery for which a paravertebral catheter is indicated based on surgeon request as well as appropriateness of location of surgical site.
* Ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnancy.
* Coagulopathy at time of evaluation or surgery.
* Infection at the site of needle insertion.
* Allergy to local anesthetic.
* Patient refusal.
* Chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption 24 hours postoperatively | first 24 hours postoperatively
  morphine equivalents of opioids in mg will be obtained from medical record

SECONDARY OUTCOMES:
Opioid consumption 48 hours postoperatively | first 48 hours postoperatively
  morphine equivalents of opioids in mg will be obtained from medical record

CONTACTS AND LOCATIONS:
Overall Officials: Elird Bojaxhi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials